CLINICAL TRIAL: NCT01309789
Title: A Phase 1 Study of Brentuximab Vedotin Administered Sequentially and Concurrently With Multi-Agent Chemotherapy as Front-Line Therapy in Patients With CD30-Positive Mature T-Cell and NK-Cell Neoplasms, Including Systemic Anaplastic Large Cell Lymphoma
Brief Title: A Phase 1 Study of Brentuximab Vedotin Given Sequentially and Combined With Multi-Agent Chemotherapy for CD30-Positive Mature T-Cell and NK-Cell Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-011; 2010-022839-11
Expanded Access: NCT01196208 (No longer available)
Record Dates: First submitted 2011-02-25; First posted 2011-03-07 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Lymphoma, Large-Cell, Anaplastic; Lymphoma, NK-cell; Lymphoma, T-cell
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Drug Therapy; Hematologic Diseases; Lymphoma; monomethyl auristatin E; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-cell; Lymphoma, NK-cell
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma; Lymphoma, T-Cell; Hematologic Diseases | interventions — Brentuximab Vedotin; Cyclophosphamide; Prednisone; Doxorubicin; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Sequential
  Interventions: Drug: brentuximab vedotin; Drug: cyclophosphamide; Drug: prednisone; Drug: doxorubicin; Drug: vincristine
- 2 (Experimental): Combination
  Interventions: Drug: brentuximab vedotin; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone
- 3 Brentuximab vedotin/CH-P (Experimental): Combination
  Interventions: Drug: brentuximab vedotin; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone

INTERVENTIONS:
Drug: brentuximab vedotin — 1.2-1.8 mg/kg IV every 3 weeks (Cycles 1-2 and if response, Cycles 9-16)
  Other Names: SGN-35
  Arms: 1
Drug: cyclophosphamide — 750 mg/m2 IV every 3 weeks (Cycles 3-8)
  Arms: 1
Drug: brentuximab vedotin — 1.2-1.8 mg/kg IV every 3 weeks (Cycles 1-6 and if response, Cycles 7-16)
  Other Names: SGN-35
  Arms: 2; 3 Brentuximab vedotin/CH-P
Drug: prednisone — 100 mg daily PO on Days 1-5 every 3 weeks (Cycles 3-8)
  Arms: 1
Drug: cyclophosphamide — 750 mg/m2 IV every 3 weeks (Cycles 1-6)
  Arms: 2; 3 Brentuximab vedotin/CH-P
Drug: doxorubicin — 50 mg/m2 IV every 3 weeks (Cycles 3-8)
  Arms: 1
Drug: doxorubicin — 50 mg/m2 IV every 3 weeks (Cycles 1-6)
  Arms: 2; 3 Brentuximab vedotin/CH-P
Drug: prednisone — 100 mg daily PO on Days 1-5 every 3 weeks (Cycles 1-6)
  Arms: 2; 3 Brentuximab vedotin/CH-P
Drug: vincristine — 1.4 mg/m2 IV every 3 weeks (Cycles 3-8)
  Arms: 1

SUMMARY:
The purpose of this study is to assess the safety profile of brentuximab vedotin sequentially and in combination with multi-agent chemotherapy in front-line treatment for CD30-positive mature T-cell and NK-cell neoplasms, including systemic anaplastic large cell lymphoma. It is a phase 1, open-label, dose escalation study in three arms designed to define the MTD, PK, immunogenicity, and anti-tumor activity of brentuximab vedotin in sequence and in combination with multi-agent front-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive CD30-positive mature T-cell and NK-cell neoplasms, including systemic anaplastic large cell lymphoma
* Measurable disease of at least 1.5 cm
* ECOG performance status less than or equal to 2

Exclusion Criteria:

* Known cerebral/meningeal disease, including history of progressive multifocal leukoencephalopathy
* Current diagnosis of primary cutaneous anaplastic large cell lymphoma, mycosis fungoides, Sezary syndrome or other primary cutaneous lymphomas; extranodal NK/T-cell lymphoma, nasal type
* History of another primary malignancy that has not been in remission for at least 3 years
* Left ventricular ejection fraction <45% or symptomatic cardiac disease, or myocardial infarction within the past 12 months
* Viral, bacterial, or fungal infection within two weeks prior to the first dose of brentuximab vedotin
* Known human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | Through 1 month after last dose

SECONDARY OUTCOMES:
Brentuximab vedotin concentration in blood | Through 1 month after last dose
Antitherapeutic antibodies in blood | Through 1 month after last dose
Best clinical response | Through 1 month after last dose
Progression-free survival | Until disease progression or study closure
Overall survival | Every 3 months until death or study closure

CONTACTS AND LOCATIONS:
Overall Officials: Dana Kennedy, PharmD, BCOP, Study Director — Seagen Inc.
Locations (11):
- United States (9):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - St. Francis Hospital, Greenville, South Carolina
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Seattle Cancer Care Alliance / University of Washington Medical Center, Seattle, Washington
- United Kingdom (2):
  - Christie Hospital NHS Foundation Trust, Manchester
  - Southampton General Hospital, Southampton

REFERENCES:
- [Result] Fanale MA, Horwitz SM, Forero-Torres A, Bartlett NL, Advani RH, Pro B, Chen RW, Davies A, Illidge T, Huebner D, Kennedy DA, Shustov AR. Brentuximab vedotin in the front-line treatment of patients with CD30+ peripheral T-cell lymphomas: results of a phase I study. J Clin Oncol. 2014 Oct 1;32(28):3137-43. doi: 10.1200/JCO.2013.54.2456. Epub 2014 Aug 18. PMID 25135998
- [Derived] Fanale MA, Horwitz SM, Forero-Torres A, Bartlett NL, Advani RH, Pro B, Chen RW, Davies A, Illidge T, Uttarwar M, Lee SY, Ren H, Kennedy DA, Shustov AR. Five-year outcomes for frontline brentuximab vedotin with CHP for CD30-expressing peripheral T-cell lymphomas. Blood. 2018 May 10;131(19):2120-2124. doi: 10.1182/blood-2017-12-821009. Epub 2018 Mar 5. PMID 29507077